CLINICAL TRIAL: NCT06048107
Title: Teniposide Incorporating Bu/Cy Conditioning Regimen Followed by HSCT for HLH With Central Nervous System Involvement: a Prospective Single-arm Clinical Study
Brief Title: Teniposide Incorporating Bu/Cy Conditioning Regimen for HLH With Central Nervous System Involvemen
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BFH20230727002/BFHHZS20230169
Record Dates: First submitted 2023-09-15; First posted 2023-09-21 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-09

CONDITIONS: HLH
MeSH Terms: interventions — Teniposide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- a prospective single-arm clinical study (Experimental)
  Interventions: Drug: Teniposide

INTERVENTIONS:
Drug: Teniposide — Teniposide is semisynthetic analogues of podophyllotoxin, and they are used in the treatment of leukemia, lymphoma, and certain sorts of solid tumors.In addition, tiniposide has central permeability and is commonly used in the treatment of central nervous system tumors.
  Other Names: VM-26

SUMMARY:
Hemophagocytic lymphohistiocytosis (HLH) is a highly inflammatory disease involving cytokine storms and is characterised by rapid progression and high mortality. There are no uniform clinical criteria for the diagnosis of CNS-HLH.And there is still a lack of international consensus on the treatment for CNS-HLH. Following allogeneic HSCT after HLH induction therapy is recommended for CNS-HLH. One of the major factors influencing the transplantation effect is conditioning. Therefore, we conduct a prospective clinical study to explore the efficacy and safety of Teniposide incorporating Bu/Cy conditioning regimen followed by allogeneic hematopoietic stem cell transplantation for HLH with central nervous system involvement.

DETAILED DESCRIPTION:
Hemophagocytic lymphohistiocytosis (HLH) is a highly inflammatory disease involving cytokine storms and is characterised by rapid progression and high mortality. HLH with central nervous system involvement (CNS-HLH) is a type of inflammatory factor storm that affects the blood-brain barrier and further infiltrates brain tissue, causing patients to exhibit corresponding neurological and/or psychiatric symptoms. It can be the first symptom of HLH or occur in the later stages of HLH, and can be an independent symptom or accompanied by other symptoms. In recent years, with the deepening of research on HLH, CNS-HLH has gradually received attention and is often associated with poor prognosis. There are no uniform clinical criteria for the diagnosis of CNS-HLH. And there is still a lack of international consensus on the treatment for CNS-HLH. Following allogeneic HSCT after HLH induction therapy is recommended for CNS-HLH. One of the major factors influencing the transplantation effect is conditioning. Therefore, we conduct a prospective clinical study to explore the efficacy and safety of Teniposide incorporating Bu/Cy conditioning regimen followed by allogeneic hematopoietic stem cell transplantation for CNS-HLH.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as HLH according to HLH-04 diagnostic criteria.
2. The indications for the presence of allogeneic hematopoietic stem cell transplantation (allo HSCT) include: I. Primary HLH; II. Refractory/recurrent HLH; III. Severe CNS-HLH.
3. According to the different causes of HLH, meeting the following conditions is defined as CNS-HLH.

   I. Definition of CNS-HLH in EBV-HLH: a significant increase of EBV-DNA copies/ml in peripheral blood or tissue or EBER(+) in tissue specimens or peripheral blood. Meanwhile cerebrospinal fluid EBV-DNA ≥5×10^2 copies/ml.

   II.Definition of CNS-HLH in primary HLH: Nervous system symptom/sign or cerebrospinal fluid cell increase (> 5 cells/μ L) and/or cerebrospinal fluid protein abnormality (> 35mg/dL) and/or brain parenchyma or meningeal abnormality in cranial imaging during the onset or course of HLH.

   III. Definition of CNS-HLH of lymphoma-associated HLH: Cerebrospinal fluid flow cytology or brain histopathology confirmed that lymphoma involved CNS. Cerebrospinal fluid EBV-DNA ≥5×10^2 copies/ml are also defined as CNS-HLH for EBV positive lymphoma-associated HLH.
4. Estimated survival time ≥ 1 month.
5. Age 14~60# gender is not limited.
6. Total bilirubin ≤ 2 times the upper limit of normal; serum creatinine ≤normal value before study entry.
7. Serum HIV antigen or antibody negative.
8. HCV antibody negative.
9. HBsAg negative, HBcAb negative. If any of the above is positive, then HBV-DNA titer in peripheral blood is required less than 1×10^2 copies/mL before enrollment.
10. Cardiac ultrasound LVEF≥50%.
11. Women in the child-bearing period must not be pregnant as determined by a pregnancy test and must be willing to use effective contraception during the trial and for ≥ 12 months after the last dose. Pregnant and lactating women cannot participate. All male subjects accept contraception during the trial and for ≥6 months after the last dose.
12. Signed informed consent.

Exclusion Criteria:

1. Heart function above grade II (NYHA).
2. Active bleeding of the internal organs(digestive tract, lung, brain, etc.).
3. Uncontrolled infection (pulmonary infection, intestinal infection, etc.).
4. Severe mental illness.
5. Patients are unable to comply during the trial and/or follow-up phase.
6. Participate in other clinical research at the same time.

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-22 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
The clinical remission rate | 24 weeks
  The number of cases with complete response (CR) and partial response (PR) after ransplantation as a percentage of the total cases.

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Wang, Principal Investigator — Department of Hematology, Affiliated Beijing Friendship Hospital, Capital Medical University
Locations (1):
- Zhao Wang, Beijing, China